CLINICAL TRIAL: NCT07131553
Title: Utvärdering av Rullstolsskolan Drivkraft en Klinisk Studie av Ett beprövat Koncept
Brief Title: Evaluation of the Wheelchair School (Drivkraft) a Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Aleris Rehab Station, Stockholm (Unknown)
Responsible Party: Principal Investigator, Emelie Butler Forslund, Principal Investigator, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2023-06358-01
Record Dates: First submitted 2025-06-27; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Neurological Disorders; Wheelchair Mobility; Rehabilitation
Keywords: wheelchair skills; spinal cord injury; multiple sclerosis; wheelchair user
MeSH Terms: conditions — Nervous System Diseases; Spinal Cord Injuries; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group wheelchair school (Experimental): Wheelchair school, 15 half days of wheelchair training
  Interventions: Other: Wheelchair school
- Comparison group (Active Comparator): conventional rehabilitation
  Interventions: Other: Comparison group, conventional rehabilitation

INTERVENTIONS:
Other: Wheelchair school — Wheelchair skills training with pysiotherapist and peer mentor
  Arms: Intervention group wheelchair school
Other: Comparison group, conventional rehabilitation — Conventional rehabilitation at the same unit of similiar length and intensity
  Other Names: Conventional rehabilitation
  Arms: Comparison group

SUMMARY:
This project will evaluate the Wheelchair School with the Drivkraft Methodology in a clinical setting. Participants are adults with chronic neurological diagnoses. For a person requiring a wheelchair, a well-functioning, individually adapted wheelchair and good maneuvering skills are essential for an independent daily life. These factors are also crucial in reducing the risk of secondary complications and pain. The Wheelchair School was founded in the 1990s, is provided by referral and both peer mentors and physiotherapists collaborate. It includes wheelchair prescription and adjustments, individually adapted wheelchair skills training, and theoretical lessons in group during 16 half-day sessions.

The overarching aim is to evaluate the intervention Wheelchair school with the Drivkraft method, for wheelchair skills and patient safety for persons with chronic neurological diagnoses in a Swedish context. Also to evaluate the psychometric properties of the Drivkraft Manouevering Test (DWMT) for wheelchair skills.

DETAILED DESCRIPTION:
Evaluation of the Wheelchair School using the Drivkraft Methodology This study focuses on adults with permanent neurological diagnoses (e.g., multiple sclerosis -MS, spinal cord injury) who continuously use a wheelchair. Education in a group setting with peer mentors who have personal experience of using a wheelchair, alongside interaction with other participants in similar situations, can be highly beneficial. The training program includes individual wheelchair prescription and or adjustments, wheelchair technique instruction, theoretical lessons, and group training. The program consists of 16 half-day sessions with peer mentors and physiotherapists in a clinical setting.

Research questions:

Do the participants improve in the following aspects directly after, and two months after the intervention: Wheelchair skills (WST and DWMT), satisfaction during everyday activities (Wheelchair Outcome Measure [WhoM]), confidence during everyday activities (Wheelchair confidence measure [WCM]), shoulder pain (wheelchair user shoulder pain index [WUSPI],fear and concerns about falling (Falls Concern Scale[FCS]), and number of falls and fall-related injuries? Is improvement of wheelchair skills associated with higher satisfaction and confidence, as well as decreased concerns about falling during daily activities? Does DWMT have sound psychometric properties, validity and sensitivity to change compared to WST? Method Design: A prospective intervention study with a comparison group. Participants: Adults with permanent neurological diagnoses referred to the Wheelchair School at Aleris Rehab Station, Stockholm, Sweden. The active comparison group comprises individuals with similar diagnoses in the same age range participating in other programs of similar length and intensity at the same unit.

Procedure: All participants undergo a physiotherapy assessment, assessment of the wheelchair including settings and manouvering skills (DWMT, WST). Also, the participants answer patient reported outcome measures (WCM, WhOM, FCS), before, directly after the rehabilitation, and after two months. The active comparison group are assessed at the same time points with the same outcome measures. The program consists of 15 half-day training sessions, and a follow-up. Psychometric properties and validity of the DWMT will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Participant in the Drivkraft Wheelchair school at Aleris Rehab Station
* Adult with neurological diagnosis using manual wheelchair

Exclusion Criteria:

* Persons with Parkinsons Disease
* Persons with too limited Swedish language skills to fill in study forms or make a signed consent
* Persons with cognitive impairments affecting their ability to fill in study forms or make a signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Drivkraft manouevering test | baseline, post intervention and at 2 months follow-up
  Test of wheelchair skills: curbs, slalom, ramps and wheelies

SECONDARY OUTCOMES:
Wheelchair outcome measure (WhOM) | baseline, post intervention and at 2 months follow-up
  A patient-reported outcome measure. Assesses how satisfied a person is when performing three self- selected everyday activity in which they use their wheelchair. They rate importance of the activity 0 (not important)-10 (most importance) and satisfaction with the activity 0 (not satisfied at all) -10 (extremely satisfied). Importance x satisfaction are compared before and after intervention
Wheelchair Skills Test (WST) | baseline, post intervention and at 2 months follow-up
  Assesses wheelchair skills: manouvering obstacles, ramps, wheelies etc
Spinal Cord Injury Falls Concern Scale (SCI-FCS) | baseline, post intervention and at 2 months follow-up
  A patient-reported outcome measure. Concerns about falling are assessed during 16 everyday activities. The person assess concerns about falling from 1 (no concern about falling) to 4 very concerned. Max 64 points

CONTACTS AND LOCATIONS:
Locations (1):
- Aleris Rehab Station, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No
Due to Swedish law, some data might be shared upon reasonable request